CLINICAL TRIAL: NCT00926419
Title: Serological Evaluation of Chickenpox (Varicella) and Hepatitis A Vaccines Using Disposable Needle-Free Syringe Jet Injector (DSJI) Delivery
Brief Title: Serological Evaluation of Varicella and Hepatitis A Vaccines Using Injector Delivery
Acronym: InjHepAVar
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Sao Paulo General Hospital (Other)
Responsible Party: Glacus de Souza Brito, Hospital das Clínicas da Faculdade de Medicina da Universidade de São Paulo
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: CAPPesq 0911/08
Record Dates: First submitted 2009-06-19; First posted 2009-06-23 (Estimated); Last update posted 2009-06-23 (Estimated); Status verified 2009-05

CONDITIONS: Varicella; Hepatitis A
Keywords: Varicella; Hepatitis A; Vaccine; Injector; Fractional dose; Intradermal; Children
MeSH Terms: conditions — Chickenpox; Hepatitis A | interventions — Chickenpox Vaccine; Hepatitis A Vaccines

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (10):
- Varicella (1/5 dose) - ID - Injector (Experimental): Lyophilized Varicella virus vaccine, live, attenuated (Oka-strain) reconstituted in 0.5 ml, Single dose, 0.1 ml Intradermal administration with Disposable Needle-free Syringe Jet Injector
  Interventions: Biological: Varicella Vaccine
- Varicella (1/5 dose) - ID - Syringe (Experimental): Lyophilized Varicella virus vaccine, live, attenuated (Oka-strain) reconstituted in 0.5 ml, Single dose, 0.1 ml Intradermal administration with Disposable Needle Syringe
  Interventions: Biological: Varicella Vaccine
- Varicella (2/5 dose) - ID - Injector (Experimental): Lyophilized Varicella virus vaccine, live, attenuated (Oka-strain) reconstituted in 0.25 ml, Single dose, 0.1 ml Intradermal administration with Disposable Needle-free Syringe Jet Injector
  Interventions: Biological: Varicella Vaccine
- Varicella (2/5 dose) - ID - Syringe (Experimental): Lyophilized Varicella virus vaccine, live, attenuated (Oka-strain) reconstituted in 0.25 ml, Single dose, 0.1 ml Intradermal administration with Disposable Needle Syringe
  Interventions: Biological: Varicella Vaccine
- Varicella (full dose) - SC - Injector (Active Comparator): Lyophilized Varicella virus vaccine, live, attenuated (Oka-strain) reconstituted in 0.5 ml, Single dose, 0.5 ml Subcutaneous administration with Disposable Needle-free Syringe Jet Injector
  Interventions: Biological: Varicella Vaccine
- Varicella (full dose) - SC - Syringe (Active Comparator): Lyophilized Varicella virus vaccine, live, attenuated (Oka-strain) reconstituted in 0.5 ml, Single dose, 0.5 ml Subcutaneous administration with Disposable Needle Syringe
  Interventions: Biological: Varicella Vaccine
- Hepatitis A (1/5 dose) ID - Injector (Experimental): Hepatitis A virus vaccine, inactivated, Single dose, 0.1 ml Intradermal administration with Disposable Needle-free Syringe Jet Injector
  Interventions: Biological: Hepatitis A Vaccine
- Hepatitis A (1/5 dose) ID - Syringe (Experimental): Hepatitis A virus vaccine, inactivated, Single dose, 0.1 ml Intradermal administration with Disposable Needle Syringe
  Interventions: Biological: Hepatitis A Vaccine
- Hepatitis A (full dose) IM - Injector (Active Comparator): Hepatitis A virus vaccine, inactivated, Single dose, 0.5 ml Intramuscular administration with Disposable Needle-free Syringe Jet Injector
  Interventions: Biological: Hepatitis A Vaccine
- Hepatitis A (full dose) IM - Syringe (Active Comparator): Hepatitis A virus vaccine, inactivated, Single dose, 0.5 ml Intramuscular administration with Disposable Needle Syringe
  Interventions: Biological: Hepatitis A Vaccine

INTERVENTIONS:
Biological: Varicella Vaccine — Lyophilized Varicella virus vaccine, live, attenuated (Oka-strain)
  Other Names: PharmaJet
  Arms: Varicella (1/5 dose) - ID - Injector; Varicella (1/5 dose) - ID - Syringe; Varicella (2/5 dose) - ID - Injector; Varicella (2/5 dose) - ID - Syringe; Varicella (full dose) - SC - Injector; Varicella (full dose) - SC - Syringe
Biological: Hepatitis A Vaccine — Hepatitis A virus vaccine, inactivated, Single dose
  Arms: Hepatitis A (1/5 dose) ID - Injector; Hepatitis A (1/5 dose) ID - Syringe; Hepatitis A (full dose) IM - Injector; Hepatitis A (full dose) IM - Syringe

SUMMARY:
This study aims to assess immunogenicity and safety of nd influence of the delivery system (needle-free injector or syringe with needle) of fractional doses (dose sparing) of two vaccines (Varicella and Hepatitis A vaccines) in children aged 13 to 30 months.

DETAILED DESCRIPTION:
The purpose of this study is to evaluate the immunogenicity, safety and influence of the delivery system (needle-free injector or syringe with needle) of fractional doses (dose sparing) (23,3 and 43,3 PFU - plaque-forming units - of live attenuated OKA strain of Varicella-zoster virus and 100 radioimmunoassay units HAV) of chickenpox and Hepatitis A ( vaccines, intradermally administered, compared with full dose of 103,3 PFU, subcutaneously administered, in 600 primo (first) vaccinated children aged 13 to 30 months selected at random at day care centers in São Paulo. Vaccines will be tested sequentially (Varicella on day 0 and Hepatitis A on day 45). Only 400 children will be randomized again for Hepatitis A vaccine testing, the remaining 200 children will receive the regular dose of Hepatitis A vaccine without further assessment. Doses will be administered using two systems: Disposable Needle-free Syringe Jet Injector (DSJI), compared with the conventional procedure using syringes and needles. Serial blood samples will be blindly analyzed to detect antibody seroconversion. Local and systemic adverse events will be assessed according to definition established by Brighton Collaboration Group, 24 and 72 hours, 7 days, 14 days, 21 days and 45 days after each vaccination, through clinical evaluation and telephone calls.

ELIGIBILITY:
Inclusion Criteria:

* Children of both genders older than 13 months and younger than 30 months of age.
* Available for follow-up for at least 45 days at public day care centers funded by São Paulo City local government.
* Written informed consent signed by parents or legal guardians after reading and explanation

Exclusion Criteria:

* Suspect/verified diagnosis of congenital or acquired immunodeficiency syndrome (AIDS)
* Suspect/verified diagnosis of malign neoplasia
* Children on treatment with high-dose systemic corticosteroids (equivalent to prednisone 2 mg/kg/day, for two or more weeks), or immunosuppressive therapy.
* Received a vaccine with live attenuated strain of virus within less than 30 days
* Suspect/verified diagnosis of chickenpox or has already been immunized against chickenpox (varicella).
* Suspect/verified diagnosis of hypersensibility to any ingredient of the vaccine.
* One of the parents or legal guardians of the minor does not agree with the study.
* Any other circumstances that may potentially damage the minor or prevent procedures from being carried out according to evaluation of the research team.
* Child shows signs or symptoms of an active intercurrent disease (e.g. fever, rash, etc.) that may interfere with the evaluation of adverse events after immunization at the research team's discretion. In this case, the participant may be reevaluated within the following three months in order to verify eligibility.

Ages: 13 Months to 30 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 600 (Estimated)
Dates: Start 2009-06; Primary Completion 2009-11 (Estimated); Study Completion 2010-05 (Estimated)

PRIMARY OUTCOMES:
Immunogenicity: General seroconversion rate 45 days following immunization. Safety: General rate of local and systemic adverse events after immunization according to definition established by Brighton Collaboration Group | 45 days after immunization

SECONDARY OUTCOMES:
Degree and duration of local and systemic adverse events after immunization according to the Brighton Collaboration Group recommendations. | 45 days after immunization
Seroconversion rates and number of local and systemic adverse events after immunization according to delivery system (needle-free injector or syringe with needle) for each dose tested | 45 days after immunization
Actual volume administered intradermally according to the delivery system (needle-free injector or syringe with needle) for each fractional dose tested | At immunization
Participants' parents or legal guardians acceptability according to the delivery system (needle-free injector or syringe with needle) for each dose tested | 45 days after immunization
Distribution of vaccine jet evaluated through ultrasound for the needle-free injector group | 5 minutes after immunization

CONTACTS AND LOCATIONS:
Overall Officials: Glacus S Brito, MD, Principal Investigator — University of Sao Paulo
Locations (1):
- Disciplina de Immunologia Clínica e Alergia do HC- FMUSP, São Paulo, São Paulo, Brazil